CLINICAL TRIAL: NCT07149532
Title: Biofeedback Therapy Alone Versus Biofeedback Therapy With Medical Treatment for Dysfunctional Voiding in Children: A Prospective Comparative Study
Brief Title: Biofeedback Therapy Alone Versus Biofeedback Therapy With Medical Treatment for Dysfunctional Voiding in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Elmaadawy, Lecturer of Urology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR1112/2/25
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Biofeedback; Medical Treatment; Dysfunctional Voiding; Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Patients will receive the biofeedback-based pelvic floor muscle training (PFMT) alone.
  Interventions: Other: Biofeedback-based pelvic floor muscle training
- Group 2 (Experimental): Patients will receive the biofeedback-based pelvic floor muscle training (PFMT) with medical treatment.
  Interventions: Other: Biofeedback-based pelvic floor muscle training (PFMT) with medical treatment

INTERVENTIONS:
Other: Biofeedback-based pelvic floor muscle training — Patients will receive the biofeedback-based pelvic floor muscle training (PFMT) alone.
  Arms: Group 1
Other: Biofeedback-based pelvic floor muscle training (PFMT) with medical treatment — Patients will receive the biofeedback-based pelvic floor muscle training (PFMT) with medical treatment.
  Arms: Group 2

SUMMARY:
This study aims to compare the efficiency of biofeedback therapy alone versus biofeedback therapy with medical treatment for dysfunctional voiding in children.

DETAILED DESCRIPTION:
Dysfunctional voiding (DV) in children may result in lower urinary tract symptoms (LUTS), such as urgency, frequency, urinary incontinence, and difficulty in urination.

Noninvasive assessments and biofeedback-based pelvic floor muscle training (PFMT) can effectively improve LUTS and protect upper urinary tract function in children, in addition to medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 18 years old.
* Both sexes.
* Children with dysfunctional voiding.

Exclusion Criteria:

* Patients with cognitive function impairment.
* Patients who received any care for dysfunctional voiding.
* Children with known anatomical anomalies of the urinary tract.
* Children with known neurological anomalies (spinal dysraphism, multiple sclerosis, lumbar or spinal neuritis……… etc).
* Children with a history of back or lower urinary tract trauma.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 months post-procedure
  Overall response rate will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.